CLINICAL TRIAL: NCT04411602
Title: Intermediate IND Severe Illness COVID-19 CP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants due to waning pandemic.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1589349
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2021-07

CONDITIONS: Severe Acute Respiratory Syndrome; COVID
Keywords: Corona Virus; Convalescent plasma
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Severely ill patients with COVID-19 severe respiratory distress
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Convalescent Plasma (Experimental): SARS-CoV-2 convalescent plasma from approved donors will be transfused into severely ill patients with confirmed COVID-19 severe respiratory distress. Plasma will be administered on days 0, 2,4, 6 and 8.
  Interventions: Drug: SARS-CoV-2 plasma

INTERVENTIONS:
Drug: SARS-CoV-2 plasma — To determine feasibility of convalescent plasma for treating patients in the ICU with COVID-19.
  Other Names: Convalescent plasma

SUMMARY:
Beyond supportive care, there are currently no proven therapeutic options for pneumonia due to coronavirus disease (COVID-19), the infection caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Human convalescent plasma is an option for treatment of COVID-19 and will be available when sufficient numbers of people have recovered. Such persons should have high titer neutralizing immunoglobulin-containing plasma.

DETAILED DESCRIPTION:
Subjects will receive open-label screened plasma from COVID-19+ clinically resolved individuals (≥14 days post-resolution). Dosing of single or double plasma units (weight based < and > 90Kg) will be administered on days 0, 2, 4, 6, and 8 (based on plasma availability), or until futility (if either occurs before day 8) is determined by the ICU. Doses can be omitted at the discretion of the treating clinician (e.g., TRALI events are 100% donor-dependent and do not prohibit future transfusions).

The study drug is the investigational product, anti-SARS-CoV-2 convalescent plasma obtained from the American Red Cross or local plasma supply (medicDal center or city/region-wide shared blood bank) from patients identified as having recovered from COVID-19. Donors and samples will be screened for infections transmitted via transfusion (e.g. HIV, HBV, HCV, WNV, HTLV-I/II, T.cruzi, ZIKV) both through the use of the uniform donor questionnaire and FDA mandated blood donor screening tests. Plasma will be collected using apheresis technology or whole blood collection in accordance with standard FDA and blood bank protocols.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed COVID-19
* Severe or Immediately life threatening COVID-19
* Dyspnea
* Respiratory frequency > 30/minute
* Blood oxygen saturation <93%
* Life-threatening disease is defined as the following
* Respiratory Failure.
* Septic shock, and/or,
* Multiple organ dysfunction or failure.

Exclusion Criteria:

* Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products).
* Other documented uncontrolled infection.
* Severe DIC needing factor replacement, FFP, cryoprecipitate.
* On dialysis.
* Active intracranial bleeding.
* Clinically significant myocardial ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Transfusion of patients in the ICU with convalescent plasma for COVID-19-induced respiratory failure. | Track patient progress for 28 days post initial convalescent dose.
  Identification of patient population in ICU that are in acute respiratory failure due to COVID-19 and transfuse with convalescent plasma

SECONDARY OUTCOMES:
Ventilatory free days | Track patient progress for 28 days post initial convalescent dose.
  Measure reduction in ventilator use and/or changes in mechanical ventilator parameters
Patient mortality (including death from any cause) | Track patient progress for 28 days post initial convalescent dose.
  Measure length of stay from the time of admission to the hospital and subsequent admission to the ICU. Document resolution of COVID-19 infection or alternatively patient death.

CONTACTS AND LOCATIONS:
Overall Officials: Shukri David, MD, Principal Investigator — Ascension Providence Hospital, Southfield Campus; Debra J Levan, DO, Principal Investigator — Ascension Macomb-Oakland Hospital, Warren Campus
Locations (3):
- United States (3):
  - Ascension Providence Hospital, Novi Campus, Novi, Michigan
  - Ascension Providence Hospital, Southfield Campus, Southfield, Michigan
  - Ascension Macomb-Oakland Hospital, Warren Campus, Warren, Michigan

REFERENCES:
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Casadevall A, Pirofski LA. Antibody-mediated regulation of cellular immunity and the inflammatory response. Trends Immunol. 2003 Sep;24(9):474-8. doi: 10.1016/s1471-4906(03)00228-x. No abstract available. PMID 12967670
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] van Erp EA, Luytjes W, Ferwerda G, van Kasteren PB. Fc-Mediated Antibody Effector Functions During Respiratory Syncytial Virus Infection and Disease. Front Immunol. 2019 Mar 22;10:548. doi: 10.3389/fimmu.2019.00548. eCollection 2019. PMID 30967872
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809